CLINICAL TRIAL: NCT04069936
Title: A Phase 2a, Open-Label, Multi-Center Study to Assess the Efficacy and Safety of Marrow Infiltrating Lymphocytes - Non-Small Cell Lung Cancer (MILs™ - NSCLC) Alone or in Combination With Nivolumab With or Without Tadalafil in Subjects With Locally Advanced and Unresectable or Metastatic NSCLC Previously Treated With Anti-PD-1
Brief Title: Marrow Infiltrating Lymphocytes - Non-Small Cell Lung Cancer (MILs™ - NSCLC) Alone or in Combination With Nivolumab With or Without Tadalafil in Locally Advanced and Unresectable or Metastatic NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Resourcing
Sponsor: WindMIL Therapeutics (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLN-P18001
Record Dates: First submitted 2019-08-16; First posted 2019-08-28 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer; Lung Cancer Metastatic; Lung Cancer, Non-small Cell; Non Small Cell Lung Cancer Metastatic; NSCLC; Non-small Cell Lung Cancer; Non-small Cell Lung Cancer Metastatic
Keywords: metastatic; locally advanced; lung cancer; non-small cell lung cancer; unresectable; NSCLC; cell therapy; autologous cell therapy; adoptive cell therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis | interventions — Nivolumab; Tadalafil

STUDY DESIGN:
Intervention Model Description: In Part 1, approximately 3-6 subjects will be treated with MILs™ - NSCLC alone. Following Part 1, approximately 20 subjects will be treated with MILs™ - NSCLC plus nivolumab with or without tadalafil.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MILs™ - NSCLC plus nivolumab with or without tadalafil (Experimental): Locally advanced and unresectable and metastatic NSCLC subjects previously treated with anti-programmed cell death-1 (PD-1) will be treated with MILs™ - NSCLC plus nivolumab with or without tadalafil.
  Interventions: Biological: MILs™ - NSCLC; Biological: nivolumab; Drug: tadalafil

INTERVENTIONS:
Biological: MILs™ - NSCLC — To evaluate the safety of MILs™ - NSCLC alone in subjects with locally advanced and unresectable or metastatic NSCLC
  Other Names: Marrow Infiltrating Lymphocytes
Biological: nivolumab — To evaluate the efficacy of MILs™ - NSCLC in combination with nivolumab in subjects with locally advanced and unresectable or metastatic NSCLC
Drug: tadalafil — To evaluate the efficacy of MILs™ - NSCLC in combination with nivolumab with or without tadalafil in subjects with locally advanced and unresectable or metastatic NSCLC

SUMMARY:
The purpose of this study is to determine the safety and efficacy of MILs™ - NSCLC alone and in combination with nivolumab with or without tadalafil in subjects with locally advanced and unresectable or metastatic NSCLC who are refractory or relapsing to a PD-1 containing regimen.

DETAILED DESCRIPTION:
This study will examine the safety and efficacy of Marrow Infiltrating Lymphocytes-Non-Small Cell Lung Cancer (MILs™ - NSCLC) combined with nivolumab with or without tadalafil in subjects with locally advanced and unresectable and metastatic NSCLC who were refractory to, or have relapsed on, an anti-PD-1 containing regimen. MILs™ - NSCLC are an adoptive cell therapy product derived via the activation and expansion of bone marrow T cells. Subjects will have bone marrow harvested during the Screening Period which will be used to manufacture the MILs™ - NSCLC. The MILs™ - NSCLC will then be administered on Day 0. Nivolumab will be administered on Day 1 and will continue every four weeks until treatment discontinuation. Tadalafil will be administered on Day 1 and will continue daily until treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
2. Locally advanced and unresectable, or metastatic NSCLC.
3. Histologically or cytologically confirmed, either squamous or non-squamous NSCLC.
4. Measurable disease as per RECIST 1.1
5. Willingness to undergo bone marrow aspiration (BMA).
6. No more than one treatment regimen following an anti-PD-1 antibody containing treatment regimen prior to BMA collection.

   a. Subjects may have BMA collected while on an anti-PD-1 antibody containing treatment regimen or while on a treatment regimen immediately following an anti-PD-1 antibody containing treatment regimen.
7. BMA may be collected while on an anti-PD-1 antibody containing treatment regimen or while on a treatment regimen immediately following an anti-PD-1 antibody containing treatment regimen. However, the subjects must have radiographic evidence of disease progression prior to lymphodepletion.
8. ≥ 21 days have lapsed since last cytotoxic chemotherapy treatment prior to collection of the BMA.
9. Previous treatment with the appropriate targeted therapy if the subject has known EGFR/ALK/ROS1 rearrangements.
10. Willingness to provide a fresh tumor biopsy during Screening Period or formalin-fixed, paraffin-embedded tissue collected at the time of most recent relapse. Note: Archival tissue regardless of biopsy date may be considered.
11. Adequate renal, hepatic and bone marrow function defined as total bilirubin </= 1.5 x ULN (except for subjects with Gilbert's disease ≤ 3.0 x ULN with direct bilirubin </= 1.5 x ULN ). Aminotransferase (AST) / Alanine Aminotransferase (ALT) </= 3.0 X ULN (subjects with liver involvement will be allowed </= 5.0 X ULN). Serum creatinine </= 1.5 x ULN; if serum creatinine is 1.5 to 2.0 × ULN, then the creatinine clearance (calculated using the Cockcroft-Gault formula or measured) must be ≥ 40 mL/min. Lymphocyte >/= 0.7 x 10^9/L. ANC >/= 1.5 x 10^9/L. Platelets >/= 100 × 10^9/L. WBC >/= 2.0 ×10^9/L. Hemoglobin > 9.0 g/dL.
12. Women of childbearing potential and male subjects (even if they are surgically sterilized or had a vasectomy) and their partners must agree to abstain or to use an effective form of birth control during the study for at least 6 months following administration of the last dose of lymphodepletion or for at least 5 months following the last dose of nivolumab for females and 7 months for males, whichever is longer. In addition, male subjects must not donate sperm during this period.
13. Capable of giving and has provided a signed ICF, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

1. Insufficient activation/expansion of T cells or other problems with the subject's MILs™ - NSCLC product which would prohibit administration.
2. Major surgical procedure within 7 days of the first dose of lymphodepletion treatment.
3. Prior malignancy active within the previous 3 years from date of BMA collection except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
4. Subjects with symptomatic uncontrolled brain metastases requiring treatment with steroids or anti-seizure medications within 28 days prior to the BMA are excluded. However, participants with brain metastases that have been previously treated and are stable on subsequent scan(s) are allowed and subjects with untreated possible brain metastases that are new at the time of screening and are < 1 cm and asymptomatic are allowed. Subjects with asymptomatic untreated CNS disease may undergo BMA prior to treatment of such disease.
5. Infection requiring treatment with intravenous antibiotics, antifungal, or antiviral agents within 7 days prior to the BMA.
6. Presence of an autoimmune disease requiring active systemic treatment.
7. Clinically significant, uncontrolled cardiovascular disease, including congestive heart failure Grade III or IV according to the New York Heart Association classification, myocardial infarction or unstable angina within the previous 6 months prior to BMA collection.
8. Known diagnosis of human immunodeficiency virus (HIV) or active viral hepatitis.
9. Administration of neutrophil growth factor support within 14 days prior to the BMA.
10. Use of systemic corticosteroids (glucocorticoids) for greater than one day within 28 days prior to the BMA.
11. Planned use of systemic corticosteroids (glucocorticoids) for greater than one day within 28 days prior to MILs™ - NSCLC administration.
12. Prior radiation to both sides of the pelvis. Prior radiation to one side of the pelvis is permitted as long as the other side of the pelvis.
13. Subjects with history of life-threatening toxicity related to prior immune therapy except those that are unlikely to re-occur with standard countermeasures.
14. Receipt of live attenuated vaccine within 30 days of planned Day 0.
15. History of allergy or hypersensitivity to MILs™-NSCLC, cyclophosphamide, fludarabine, nivolumab, tadalafil or their components.
16. Pregnant or lactating females.
17. Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's opinion, could affect the safety of the subject or impair the assessment of study results.
18. Unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0 | From ICF through 100 days after the last dose of study treatment
  Incidence, intensity, and type of AE
Serious Adverse Events per NCI-CTCAE version 5.0 | From ICF through 100 days after the last dose of study treatment
  Incidence, intensity, and type of SAE
Overall Response Rate (ORR) of MILs™ - NSCLC in combination with nivolumab with or without tadalafil | 24 months
  Proportion of subjects with reduction in tumor burden of a predefined amount per RECIST 1.1

SECONDARY OUTCOMES:
Duration of response | up to 5 years after treatment discontinuation
  Duration from first documented evidence of CR or PR until the first documented evidence of PD or death due to any cause, whichever occurs first
Disease control rate | up to 5 years after treatment discontinuation
  Proportion of subjects in the efficacy population who achieve an Investigator-assessed confirmed CR, PR, or SD per RECIST 1.1
Progression-free survival | up to 5 years after treatment discontinuation
  Date of first the administration of MILs™ - NSCLC until documented PD or death due to any cause, whichever occurs first
Overall survival | up to 5 years after treatment discontinuation
  Duration from the date of administration of MILs™ - NSCLC until death due to any cause
Overall Response Rate (ORR) of MILs™ - NSCLC | 24 months
  Proportion of subjects with reduction in tumor burden of a predefined amount per RECIST 1.1
Safety of MILs™ - NSCLC alone and in combination with nivolumab with or without tadalafil as assessed by vital signs (pulse rate) | From ICF through 100 days after the last dose of study treatment
  Pulse rate in beats/minute
Safety of MILs™ - NSCLC alone and in combination with nivolumab with or without tadalafil as assessed by vital signs (weight) | From ICF through 100 days after the last dose of study treatment
  Weight in pounds
Safety of MILs™ - NSCLC alone and in combination with nivolumab with or without tadalafil as assessed by vital signs (blood pressure) | From ICF through 100 days after the last dose of study treatment
  Systolic and diastolic blood pressure in mmHg
Safety of MILs™ - NSCLC alone and in combination with nivolumab with or without tadalafil as assessed by vital signs (respiratory rate) | From ICF through 100 days after the last dose of study treatment
  Respiratory rate in breaths/minute
Safety of MILs™ - NSCLC alone and in combination with nivolumab with or without tadalafil as assessed by vital signs (temperature) | From ICF through 100 days after the last dose of study treatment
  Termperature in Fahrenheit
Safety of MILs™ - NSCLC alone and in combination with nivo. with or w/o tadalafil by liver function (ALT/AST (U/L), albumin (g/dL), tot. bilirubin (mg/dL)), kidney function (creatinine (mg/dL) and endocrine function (T3 free and T4 free (ng/dL)) | From ICF through 100 days after the last dose of study treatment
  Clinical chemistry results will be summarized and changes from baseline provided
Safety of MILs™ - NSCLC alone and in combination with nivolumab with or without tadalafil by cell count (e.g. RBC (10^6/uL), WBC (10^3/uL), absolute cell count (10^3/uL), Hct (%) and Hgb (g/dL) | From ICF through 100 days after the last dose of study treatment
  Hematology results will be summarized and changes from baseline provided
Safety of MILs™ - NSCLC alone and in combination with nivolumab with or without tadalafil as assessed by APTT (seconds), fibrinogen (mg/dL), INR and protime (seconds) | From ICF through 100 days after the last dose of study treatment
  Coagulation results will be summarized in data listings
Safety of MILs™ - NSCLC alone and in combination with nivolumab with or without tadalafil as assessed by urine appearance, color, pH, specific gravity and presence of blood, bilirubin, glucose, ketone, leukocyte esterase, nitrite, protein, urobilinogen | From ICF through 100 days after the last dose of study treatment
  Urinalysis results will be summarized in data listings
Safety of MILs™ - NSCLC alone and in combination with nivolumab with or without tadalafil by electrocardiograms (ECGs) assessed by Investigators as normal, abnormal clinically significant or abnormal not clinically significant | From ICF through 100 days after the last dose of study treatment
  ECGs results will be summarized and changes from baseline provided
Safety of MILs™ - NSCLC alone and in combination with nivolumab with or without tadalafil by physical examination with abnormalities reported as adverse events | From ICF through 100 days after the last dose of study treatment
  Physical examinations will be performed by the Investigators and any new clinically significant or changes in medical conditions will be reported as adverse events

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - City of Hope, Duarte, California
  - University of California - Los Angeles, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Karmanos Cancer Center, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No